CLINICAL TRIAL: NCT05977218
Title: DIgitAl diabeTES Treatment - the Healthy Eating, heaLthy Patients Trial
Acronym: DIATEST-HELP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Lana Hebib, Principal investigator, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: DIATEST-HELP
Record Dates: First submitted 2023-07-06; First posted 2023-08-04 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Type 2 Diabetes
Keywords: Diet; Mobile health; HbA1c
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Access to the 'DiabetesSwitch' filter of the FoodSwitch app when grocery shopping during 26 weeks, in addition to standard written dietary advice
  Interventions: Other: FoodSwitch
- Control (No Intervention): Access to standard written dietary advice

INTERVENTIONS:
Other: FoodSwitch — Access to the 'DiabetesSwitch' filter of the FoodSwitch app when grocery shopping. When a packaged food item bar code is scanned, the FoodSwitch app will show an interpretive nutritional information score for the scanned product and recommend alternate healthier food options in the same category.
  Arms: Intervention

SUMMARY:
This randomized controlled trial will assess the impact of the FoodSwitch mobile app, which provides interpretive front-of-pack labelling via barcode scanning, in 900 Swedish adults with type 2 diabetes. Participants will be randomized to app + standard advice or standard advice alone. The primary outcome is change in HbA1c at 6 months; secondary outcomes include anthropometrics, quality of life, medication use, hospitalizations, and mortality.

DETAILED DESCRIPTION:
A healthy diet improves glycaemic control and reduces cardiovascular risk in type 2 diabetes (T2D), but access to dietitians is limited. Unlike several countries, Sweden has not implemented interpretive front-of-pack labelling. Smartphone applications may offer an alternative. This trial evaluates the dietary and clinical impact of FoodSwitch, a mobile app providing interpretive labelling to Swedish adults with T2D. Nine hundred individuals with T2D for ≥2 years who regularly shop for groceries will be recruited via general practices and community advertisements and randomized to receive access to FoodSwitch plus standard written dietary advice, or standard written dietary advice only. The primary outcome is change in self-measured glycated haemoglobin (HbA1c) after 6 months. Secondary outcomes include waist circumference, body weight, quality of life, dietary self-efficacy, medication use, hospitalizations, and all-cause mortality. Exploratory outcomes include omics analyses.

ELIGIBILITY:
Inclusion criteria:

* Age between 18 and 75 years
* Self-reported type 2 diabetes with a duration of ≥2 years
* Regularly grocery shopping

Exclusion criteria:

* No access to BankID (a digital identification system commonly used in Sweden)
* Failure to complete eligibility screening and run-in periods

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean HbA1c | Change from baseline at week 26
  Mean glycated haemoglobin

SECONDARY OUTCOMES:
Self-measured waist circumference (cm) | Change from baseline at week 26
  Self-measured waist circumference (cm)
Self-reported quality of life | Change from baseline at week 26
  Self-reported quality of life - questionnaire
Self-measured body weight (kg) | Change from baseline at week 26
  Self-measured body weight (kg)
Registry-based data on medication use, hospitalizations, outpatient visits, and diabetes complications | Change from baseline at week 26
  Registry-based data on medication use, hospitalizations, outpatient visits, and diabetes complications
Self-reported dietary self-efficacy | Change from baseline at week 26
  Self-reported dietary self-efficacy
Difference in all-cause mortality | Change from baseline at week 26
  Difference in all-cause mortality

OTHER OUTCOMES:
Dietary effects on proteomics and metabolomics | Change from baseline at week 26
  Dietary effects on proteomics and metabolomics

CONTACTS AND LOCATIONS:
Overall Officials: Karin Rådholm, MD, PhD, Study Director — Linkoeping University
Locations (1):
- Linköping University, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: After publication in a peer-reviewed journal and for the period of time for which local archive regulations stipulate.
Access Criteria: To be determined on a case by case basis.

REFERENCES:
- [Derived] Af Geijerstam P, Johansson E, Fagerstam S, Wu JH, Ghafouri B, Karlsson K, Hebib L, Kastbom L, Wennberg P, Gustafson Hedov E, Storgards M, Sundstrom J, Radholm K. Effect of the FoodSwitch application on type 2 diabetes in Sweden: a study protocol for the randomised controlled DIgitAl diabeTES Treatment - the Healthy Eating, heaLthy Patients trial (DIATEST-HELP). BMJ Open. 2025 Nov 16;15(11):e110141. doi: 10.1136/bmjopen-2025-110141. PMID 41248424